### **Research Study Informed Consent Document**

**Study Title for Participants:** Testing the use of fulvestrant and binimetinib targeted treatment for nfl mutation in hormone receptor-positive metastatic breast cancer

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Molecular Analysis for Combination Therapy Choice (ComboMATCH)

A ComboMATCH Treatment Trial: Protocol EAY191-N2: Phase 2 Trial of Fulvestrant and Binimetinib in Patients with Hormone Receptor-Positive Metastatic Breast Cancer with Inactivating or Inferred Inactivating NF1 Alterations (NCT05554354)

### **Overview and Key Information**

# What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have breast cancer that is hormone receptor positive and has spread (metastasized) outside your breast, and your cancer has a change in the gene called the NF1 gene.

# Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

# Why is this study being done?

Please know that your eligibility for this trial may have been determined in part on the basis of a laboratory-developed test that has not been reviewed or approved by the FDA.

This study is being done to answer the following questions:

If you have never received fulvestrant (fulvestrant-naïve), can your breast cancer be stabilized and the time that you live with your breast cancer be lengthened by adding binimetinib to the usual drug fulvestrant? If you have received fulvestrant (fulvestrant exposed), has your breast cancer shrunk within 4 months of starting treatment with binimetinib added to the usual drug fulvestrant?

Protocol Version Date: 02/12/2024 

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your breast cancer that is hormone receptor-positive and has metastasized. The usual approach is defined as care most people get for hormone receptor-positive metastatic breast cancer.

# What is the usual approach to my hormone receptor-positive breast cancer that has metastasized?

There is currently no agreed upon approach for treating cancers with the genetic change that you have (NF1). People who are not in a study are usually treated with hormonal therapy. Sometimes combinations of these are used. Treatments are generally continued until the disease gets worse or side effects become too severe. Your doctor can explain which treatment may be best for you. These treatments can reduce symptoms and may stop the tumor from growing for a few months or more. The usual approach is proven to help patients with your health condition live longer.

# What are my choices if I decide not take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

# What will happen if I decide to take part in this study?

If you decide to take part in this study, you will either get the study drugs fulvestrant and binimetinib or fulvestrant alone if you are fulvestrant-naive. You will get the study drugs fulvestrant and binimetinib if you are fulvestrant-exposed. Treatment will continue until your disease gets worse, or the side effects become too severe, or you decide to stop the therapy.

After you have completed fulvestrant and binimetinib or fulvestrant alone, your doctor and study team will continue to watch you for side effects, until your disease gets worse or the side effects become too severe. They will check you every 6 months for up to 5 years. This will be done at a visit to your study doctor. You will be in this study for up to 5 years from the time you join the study.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the fulvestrant and binimetinib may not be as good as the usual approach for your cancer at stabilizing your cancer if you are fulvestrant-naïve or of shrinking your breast cancer if you are fulvestrant-exposed.


There is also a risk that you could have side effects from the fulvestrant and binimetinib. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that study doctors know about are:

- Visual disturbances
- Diarrhea, nausea, vomiting
- Swelling of the body
- Tiredness
- Acne, rash
- Cough
- Infection, especially when white blood cell count is low
- Anemia which may require transfusion
- Bruising, bleeding
- Constipation, loss of appetite
- Pain
- Flushing
- Headache

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is evidence that the treatment with binimetinib and fulvestrant is effective in stabilizing your type of cancer if you are fulvestrant-naïve or shrinking your type of cancer if you are fulvestrant-exposed. It is not possible to know now if binimetinib and fulvestrant will extend how long you live with cancer and not have it get worse compared to the usual approach. This study will help the study doctors learn things that may help people in the future.

# If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. This may mean slowly stopping the study drugs so that there is not a sudden unsafe change and risk to your health. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

# Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.


• The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (NRG Oncology). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

# What is the purpose of this study?

The purpose of this study is to compare the usual treatment alone (fulvestrant) to using binimetinib plus the usual treatment in patients whose cancer has an NF1 genetic change, and they have not received fulvestrant. The addition of binimetinib to the usual treatment could stabilize cancer. For patients who have received fulvestrant before joining the study, the study will test if adding binimetinib to fulvestrant in these patients whose cancer has an NF1 genetic change could shrink the breast cancer. But, it could also cause side effects, which are described in the risks section below.

This study will help the study doctors find out if this different approach is better, the same, or worse than the usual approach. To decide if it is better, the study doctors will be looking to see if the binimetinib lengthens the time during and after the treatment of your cancer that you live with your cancer and it is stable, or if your cancer shrinks, compared to the usual approach.

Binimetinib is already approved by the FDA for use in skin cancer. There will be about 95 people taking part in this study.

# What are the study groups?

This study has two study groups.

# • Group 1 (Patients who have never received fulvestrant)

If you are in this group, you will get the usual drug fulvestrant and the study drug binimetinib or the usual drug fulvestrant.

- If you are in Arm A, you will get fulvestrant and binimetinib. You will get fulvestrant intramuscularly (IM injection) on days 1 and 15 during the first cycle and on day 1 of each 28-day cycle afterwards. Binimetinib is a pill you take by mouth twice a day (morning and evening) on days 1 through 28 of each cycle beginning on Cycle 1, Day 15. Each cycle lasts 28 days. You will get fulvestrant and binimetinib as long as your cancer responds to the drugs and as long as your doctor thinks it is safe to keep you on them.
- If you are in Arm B, you will get fulvestrant intramuscularly (IM injection) on days 1 and 15 during the first cycle and on day 1 of each 28-day cycle afterwards. You will get fulvestrant as long as your cancer responds to the drugs and as long as your doctor thinks it is safe to keep you on them. If your cancer starts to grow while you are receiving fulvestrant alone, you will be asked to join Group 2 and to agree to receive fulvestrant and binimetinib.

There will be about 70 people in this group.


#### • Group 2 (Patients who previously received fulvestrant)

If you are in this group, you will get the usual drug fulvestrant. You will also get the study drug binimetinib. You will get fulvestrant intramuscularly (IM injection) on days 1 and 15 during the first cycle and on day 1 of each 28-day cycle afterwards. You will also take binimetinib, which is a pill you take by mouth twice a day (morning and evening), on days 1 through 28 of each cycle beginning on Cycle 1, Day 15. Each cycle lasts 28 days. You will get fulvestrant and binimetinib as long as your cancer responds to the drugs and as long as your doctor thinks it is safe to keep you on them.

There will be about 16 to 25 people in this group.

We will use a computer to assign you to one of the study groups. This process is called "randomization." It means that your doctor will not choose and you cannot choose which study group you are in. You will be put into a group by chance. You will have an equal chance of being in Arm A or Arm B if you are in Group 1. If you are in Group 2, all participants will receive the same study drugs.

Another way to find out what will happen to you during this study is to read the chart below. Start reading from the left and read across to the right, following the arrows.

**Group 1 (Patients who have never received fulvestrant)** 



<sup>\*</sup> If your cancer starts to grow while you are receiving fulvestrant alone, (Arm B), you will be asked to join Group 2 and to agree to receive fulvestrant and binimetinib.


Protocol Version Date: 02/12/2024 EAY191-N2

**Group 2 (Patients who previously received fulvestrant)** 



# What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are tests that will be done for research purposes only.

If you have biopsiable disease and a biopsy can be done with minimal risk, you will have to have a biopsy. The study biopsy takes small pieces of cancer tissue from your body. If you do not have biopsiable disease or a biopsy would not be minimal risk, you will need to have tumor tissue available from a recent biopsy. You will also have a special blood sample for the study before you begin study drug.

After you join the study and you are going to receive binimetinib, you may need to have a test that checks how well your heart is functioning if you have not already had the test. If the result is too low, you will not be able to receive study treatment. If you have had the test done within 12 weeks before starting binimetinib, it does not need to be repeated.

The cancer tissue will be used to look at why a drug may work for you or why you your tumor may not respond to a drug. Genetic tests will be performed on the submitted tissue and blood. The tissue and blood will be sent to the central ComboMATCH laboratories to see whether the ComboMATCH test results are the same as the results from the ComboMATCH-designated lab.

You and your study doctor will not get the results of this testing. If you agree to take part in the study, you may need to sign a separate consent form for the study biopsy at the hospital or clinic where the biopsy is done.

# What risks can I expect from taking part in this study?

#### General Risks

If you choose to take part in this study, there is a risk that the binimetinib and fulvestrant may not be as good as the usual approach for stabilizing your cancer.


You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The drugs used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 30 days after you complete binimetinib and for 12 months after you complete fulvestrant.

This study will use a sample of your tissue. Generally, your hospital will keep some of your tissue. This tissue may be used to help treat your cancer in the future. Because this study will need to use some of this tissue, there is a small risk that it could be used up.

#### **Biopsy Risks**

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection can occur. If your cancer starts to grow while you are receiving fulvestrant alone and you join Group 2, you will have another biopsy. The risks of another biopsy are the same as the risks already listed. You may sign a separate consent form for the study biopsy that describes the risks in more detail.

If there is any leftover specimen that may possibly be stored for biobanking, this will be discussed in the section under "Optional studies".

#### Risks of Blood Draw

The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.

#### **Side Effect Risks**

The study drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drugs.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.


#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

**Study Group 1 and Group 2:** Possible side effects of binimetinib and fulvestrant are listed in the tables below.

#### Possible Side Effects of Binimetinib (CAEPR Version 2.2, April 12, 2023)

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving binimetinib, more than 20 and up to 100 may have:

- Visual disturbances
- Diarrhea, nausea, vomiting
- Swelling of arms, legs
- Tiredness
- Acne, rash

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving binimetinib, from 4 to 20 may have:

- Anemia which may require blood transfusion
- Blurred vision
- Pain
- Constipation
- Sores in the mouth which may cause difficulty swallowing
- Fever
- Infection
- Change in heart function
- Loss of appetite
- Muscle weakness
- Dizziness
- Shortness of breath
- Hair loss, itching
- Dry skin
- Change in or loss of some or all of the finger or toenails
- A hole or tear in the skin
- High blood pressure which may cause headaches, dizziness, blurred vision
- Blood clot which may cause swelling, pain, shortness of breath

# RARE, AND SERIOUS

In 100 people receiving binimetinib, 3 or fewer may have:

- Heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- Abnormal heartbeat
- Glaucoma


#### RARE, AND SERIOUS

In 100 people receiving binimetinib, 3 or fewer may have:

- Swelling of the eye
- Visual loss
- Liver damage which may cause yellowing of eyes and skin, swelling
- Damage to the muscle which may cause muscle pain, dark red urine
- Damage to lungs which may cause shortness of breath
- Bleeding

#### Possible Side Effects of Fulvestrant (Table Version Date: August 30, 2019)

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving Fulvestrant, more than 20 and up to 100 may have:

- Cough
- Infection, especially when white blood cell count is low
- Anemia which may require transfusion
- Bruising, bleeding
- Constipation, diarrhea, nausea, vomiting, loss of appetite
- Pain
- Tiredness
- Flushing
- Headache

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Fulvestrant, from 4 to 20 may have:

- Change in the heart rhythm
- Swelling of the body
- Shortness of breath
- Blood clot which may cause swelling, pain
- Liver damage which may cause yellow eyes and skin, swelling
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat

#### RARE, AND SERIOUS

In 100 people receiving Fulvestrant, 3 or fewer may have:

• None

# **Additional Drug Risks:**

The binimetinib could interact with other drugs. Binimetinib and fulvestrant have not been studied when given together so there may be unknown risks with the use of binimetinib and fulvestrant when given together. Your study doctor will give you a clinical trial wallet card that lists the study drug that you are taking. Share this information with your family members, caregivers, other health providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.


### What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.
- Write down in your medication diary when you take binimetinib at home.

**For women:** Do not get pregnant or breastfeed while taking part in this study. **For men:** Do not father a baby while taking part in this study. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 30 days after your last dose of binimetinib and 12 months after you last dose of fulvestrant.

# What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your breast cancer. This includes:

- the cost of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the cost of getting fulvestrant ready and giving it to you.
- the test to check your heart before you start taking binimetinib.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

- The research biopsy done after enrollment to the study.
- The research studies done on the research biopsy for this study.
- The research blood samples drawn for ctDNA testing after enrollment to the study.

You or your insurance provider will not have to pay for the binimetinib while you take part in this study. You or your insurance provider will have to pay for the fulvestrant while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.


You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor and any company supporting the study drug now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.


Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

# Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) Institutional Review Board at (\*insert telephone number\*).

# Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading this optional study hope the results will help other people with cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in this optional study is your choice. You can still take part in the main study even if you say "no" to this study. There is no penalty for saying "no." You and your insurance company will not be billed for this optional study. If you sign up for, but cannot complete this study for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for the following study.


# Optional sample storage for known laboratory studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

#### Known future studies

If you choose to take part in this optional study, researchers will collect blood and tumor for research on changes in the genes in your breast cancer tumor to research why a drug may work for you or why your tumor may not respond to a drug. The researchers will also look at changes in certain biomarkers in your blood.

#### Unknown future studies

If you choose to take part in this optional study, tissue from the biopsies collected as part of the main study will be stored for future research. Storing samples for future studies is called "biobanking." The biobank is being run by ECOG/ACRIN and is supported by the NCI. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we don't know what research may be done in the future using your tissue samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes. If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.


#### What is involved in this optional sample storage?

If you agree to take part, here is what will happen next:

- 1. Your samples will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 2. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 3. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

### What are the risks in this optional sample storage?

- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone outside
  of the research study could get access to your study records or trace information in a
  database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of tracing
  information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: <a href="https://www.genome.gov/10002328/">https://www.genome.gov/10002328/</a>

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your sample and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in these optional future studies?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.


### Are there any costs or payments to these optional future studies?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

### What if I change my mind about these optional future studies?

If you decide you no longer want your samples to be used, you can call the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*), who will let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers.

#### What if I have questions about these optional future studies?

If you have questions about the use of your samples for research, contact the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*).

Please circle your answer below to show if you would or would not like to take part in the optional study:

### Blood samples for known future studies:

I agree that my blood samples and related health information may be used for the laboratory studies described above.

YES NO

### Additional biopsy for known future studies:

I agree that an additional biopsy may be done to obtain research specimens if my disease comes back or shows signs of coming back and that this sample and related health information may be used for the laboratory studies described above.

YES NO

# Samples for unknown future studies:

I agree that my samples and related health information may be kept in a biobank for use in future health research.

YES NO

#### Contact for Future Research

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

YES NO

# This is the end of the section about optional studies.


# My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

| Participant's signature |
|-------------------------------------------------------------------|
| Date of signature |
| Signature of person(s) conducting the informed consent discussion |
| Date of signature |
